CLINICAL TRIAL: NCT01187342
Title: Depression and Posttraumatic Stress Disorder in Stroke Patients: an Observational Study of Neuro-psychiatric, Cognitive, and MR-Changes Over Time After Stroke
Brief Title: Post Stroke Psychological Distress
Acronym: POSTPSYDIS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Matthias Endres, Prof. MD, Charite University, Berlin, Germany
Other Study IDs: POSTPSYDIS; 4-026-08 (Other: Ethics Committee Charité)
Record Dates: First submitted 2010-07-01; First posted 2010-08-24 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-striatal lesion group: acute ischemic Stroke in MCA territory of 10-100 cm³ with sparing of striatocapsular structures
- Striatal lesion group: acute ischemic stroke in MCA/AchA territory with involvement of at least 125 mm³ of striatocapsular structures

SUMMARY:
Neuro-psychological, cognitive and biochemical assessment matched with MR-Imaging in acute and chronic poststroke conditions.

DETAILED DESCRIPTION:
The study design relates to affective symptomatology, particularly poststroke depression and posttraumatic stress symptoms as well as to cognitive decline due to stress-related hypercortisolemia in the early phase after stroke. Extended MRI studies including a functional connectivity (fc-MRI) paradigm have been incorporated to study on subacute midbrain neurodegeneration as a possible morphological correlate of functional and clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Stroke in MCA/AchA territory of striato-capsular (at least 125mm³) or non-striatal (10-100cm³) involvement
* MR-imaging can be conducted 24-48 hours of onset
* preserved communication skills

Exclusion Criteria:

* Patients with psychiatric conditions or medication in the last 4 weeks
* severe medical conditions
* limited prognosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute ischemic stroke in MCA/AchA territory within 48 hours of onset
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
occurence of depression (GDS, SKID) | 90 days
  Geriatric Depression Scale, Structured Clinical interview for DSM-IV

SECONDARY OUTCOMES:
change in saliva cortisol | 90days
  measurement of saliva cortisol levels
change in serumcholine | 90days
  measurement of serumcholine

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Endres, MD, Study Director — Center for Stroke Research Berlin
Locations (1):
- Charité, Campus Benjamin Franklin, Dep. of Neurology, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kufner A, Rios AS, Winter B, Temuulen U, Khalil A, Grittner U, Schoner J, Akdeniz A, Lachmann U, Kronenberg G, Villringer A, Gertz K, Endres M. Neuropsychiatric changes following striatal stroke- results from the observational PostPsyDis study. Neurol Res Pract. 2025 May 12;7(1):32. doi: 10.1186/s42466-025-00390-3. PMID 40350509